CLINICAL TRIAL: NCT04792411
Title: Multi-centre, Pilot Study Evaluating the Feasibility, Acceptability, and Short-term Outcomes of a Tailored, Virtual, Home-based, Multicomponent Prehabilitation Programme in Patients Undergoing Abdominal Aortic Aneurysms (AAA) Repair.
Brief Title: Adherence and Acceptability of a Remote, Home-based, Pre-surgery Programme for Patients Undergoing Abdominal Aortic Aneurysm Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 291828
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: AAA, pre-conditioning, frailty
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation group (Experimental): This arm will be subject to at least 6 weeks of a tailored prehabilitation programme
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Multimodal, tailored prehabilitation programme

SUMMARY:
Design A multi-centre pilot study investigating the acceptability and adherence of a prehabilitation on patients requiring abdominal aortic aneurysm repair.

Setting 3 NHS Hospital Vascular Surgery Clinics in the UK.

* Imperial College Healthcare NHS Trust
* Cambridge University Hospitals NHS Trust
* Mid and South Essex NHS Trust

Patient Population Patients referred to secondary/tertiary vascular clinic for the repair of asymptomatic infrarenal Aneurysm

Intervention:

Baseline (conducted face-to-face): After providing written informed consent, participants will be provided with information about the prehabilitation programme. The following data will also be collected: baseline demographic characteristics (including age, sex and ethnicity), body mass index (BMI), medical history (including time since diagnosis), current medication, aneurysm diameter, health-related quality of life (EQ-5D-5L and EQ-VAS), smoking status and psychological wellbeing (using the Hospital Anxiety and Depression Scale; HADS) and Frailty assessments( QMortality Index, Electronic Frailty Index, Rockall score). Participants will also complete a 6-minute walking test(6MWT).

DETAILED DESCRIPTION:
Weeks 1 to 5 (conducted remotely via telephone, email or completion of an online survey):

The programme has been developed with experts in the field of sports therapy, physiotherapy and biomechanics, based on robust literature in other fields. The course plan is to start with 3 sessions every week for 6 weeks where participants would complete a tailored home exercise programme or until the expected surgical intervention. In the first week of this programme, the patient will receive three sessions with a total of 150 minutes of exercise according to UK Chief Medical Officers' Physical Activity Guidelines. After each week, we will assess patient tolerance to the exercise regime using Borg scale. The researchers will either increase or decrease exercise intensity according to their feedback. The study will also be assessing patients' preference for how and when they would like to exercise.

End of Programme (conducted remotely via telephone, email or completion of an online survey):

Participants will be contacted by a member of the study team for the reassessment of health-related quality of life, psychological wellbeing and smoking status. Participants will also be required to provide their self-reported weight. On admission for surgery, they will be assessed for frailty using frailty score assessments

Post - Operative Morbidity score(POMS) will be assessed during admission ( Day1, Day 3, Day 5, Day 7, etc) after surgery.

Discharge: (conducted either remotely or face to face):

Participants will complete a reassessment of health-related quality of life, disease-specific quality of life, psychological wellbeing and smoking status. Participants will also complete the 6-MWT.

6 weeks post-surgery (conducted remotely or face-to-face): Participants will complete a reassessment of health-related quality of life, disease-specific quality of life, psychological wellbeing and smoking status. Participants will also complete the 6-MWT.

90-days post-surgery (conducted remotely or face-to-face): Participants will complete reassessment of health-related quality of life, disease-specific quality of life, psychological wellbeing and smoking status. Participants will also complete the 6-MWT. Participants will also complete a frailty assessment score (Rockall)

Treatments Standard national and local practice will be followed for the repair of infra-renal aortic aneurysm. Patients will receive any type of repair as decided by the local Vascular Multi-Disciplinary Team.

Primary Outcome Prehabilitation Programme compliance, attendance and acceptability.

Secondary Outcomes

* In-Hospital Complication Rate - Composite of Cardiac, Respiratory, Renal, Haemorrhage, Limb Ischaemia and Cerebral Complications, as defined by National Vascular Registry
* Length of stay and readmission rates (30 days post-surgery)
* 30-day Composite Outcome: Death and Defined complication (Cardiac, respiratory, haemorrhage, limb ischaemia, renal failure)
* Change in 6-minute walk test (6-MWT) at end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge)
* Change in health-related quality of life scores (using the EuroQol five-dimensional questionnaire [EQ-5D] and visual analogue scale [EQ-VAS]) at end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge)
* Post-Operative Morbidity score (POMS)
* Change in aneurysm specific quality of life scores at end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge)
* Change in Hospital Anxiety and Depression Score (HADS) at 6-weeks post enrolment and 30 and 90-days post-surgery
* Reduction in cigarettes per day at 6-weeks post enrolment and 30 and 90-days post-surgery
* Change in weight (in kg) 6-weeks post enrolment and 30 and 90-days post-surgery

ELIGIBILITY:
Inclusion Criteria

* Adults (aged 55 years and over) who have been diagnosed with an AAA and are scheduled to undergo EVAR or open surgery (with a wait time of at least 6-weeks for surgery).
* Patients with an AAA with a diameter of 5.5cm to 7cm
* Able to write, understand and communicate in English
* Willing and able to participate in a virtual prehabilitation programme

Exclusion Criteria:

* Thoraco-Abdominal Aneurysms
* Connective tissue Vascular Disorder
* Symptomatic aneurysms
* Previous Aortic intervention
* Absolute contraindication to exercise
* Inability or unwillingness to participate in the trial
* Infrarenal AAA diameter exceeding 7.0cm
* Emergency AAA repair
* BMI below 20 kg/m2 or above 45 kg/m2

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of screening and recruitment | 18 months
  The number of participants referred at each site will be captured The number of participants eligible for screening at each site will be captured The number of participants enrolled at each site will be captured Reasons for non-participation will be captured
Feasibility of measurement tools: | 18 months
  Time taken to complete the questionnaires at each time-point The ratio of missing data from questionnaires Follow-up response rates
Adherence | at least 6 weeks ( Duration of the programme)
  Number of sessions attended The proportion of participants who complete' the 6-week programme
Acceptability of the prehabilitation programme (Patient satisfaction) | 18 months
  Patient satisfaction will be measured using questionnaires Reasons for drop-out will be captured.

SECONDARY OUTCOMES:
In-Hospital Complication Rate | Immediately after the surgery
  - Composite of Cardiac, Respiratory, Renal, Haemorrhage, Limb Ischaemia and Cerebral Complications, as defined by National Vascular Registry
30-day(After surgery) Composite Outcome | 30 days
  Incidence of Mortality Incidence of complications
Length of stay and readmission rates (30 days post-surgery) | 30 days
  Reintervention, or areadmission related to repair or other complications
Change in 6-minute walk test (6-MWT) at end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge) | 6 weeks, 3 months
  To measure the change of patient physical function
Change in health-related quality of life scores (using the EuroQol five-dimensional questionnaire [EQ-5D] and visual analogue scale [EQ-VAS]) at end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge) | 6 weeks, 3 months
  Participants quality of life measure throughout the study
Post-Operative Morbidity score (POMS) | Immediately after surgery
  To measure post operative complications and it's impact on participants
Change in aneurysm specific quality of life scores at end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge) | 6 weeks, 3 months
  Participants quality of life measure related to aneurysm repair throughout the study
Change in Hospital Anxiety and Depression Score (HADS) end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge) | 6 weeks, 3 months
  Participants anxiety and depression score change throughout the study 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
Change in cigarettes usage per day | 6 weeks, 3 months
  Difference in cigarettes usage at different phases of the study
Change in weight (in kg) end of programme, Discharge, 6-weeks (Post discharge) and 3 months (Post Discharge) | 6 weeks, 3 months
  Measure weight change

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Study Chair — Imperial College NHS Trust; Tristan Lane, Principal Investigator — Cambridge University Hospitals NHS Trust; Ankur Thapar, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No